CLINICAL TRIAL: NCT02431195
Title: Analysis of Changes in Eating Behaviors and Physical Activity on Post Bariatric Surgery Patients and Their Family Members : Comparison Between Men and Women
Brief Title: Analysis of Changes in Eating Habits on Post Bariatric Surgery Patients and Their Family Members
Acronym: SOCIOB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 13SCW-SOCIOB
Record Dates: First submitted 2015-03-17; First posted 2015-04-30 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Bariatric Surgery
Keywords: obesity; bariatric surgery; physical activity; eating habits
MeSH Terms: conditions — Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to identify changes in eating behaviors and physical activity in patients after bariatric surgery and their family members living in same household: children aged between 11-17 years, spouse, parents, cohabitee or partner in a civil union.

DETAILED DESCRIPTION:
As secondary objectives, the study aims to:

* Describe the sociodemographic and clinical characteristics of post bariatric surgery patients.
* Assess changes in quality of life of the post-surgery patients.
* Explain changes of post-surgery in eating behavior and activity varied according to gender
* Explain changes of post-surgery in eating behavior and activity varied according to socio-economic conditions
* Explain changes of post-surgery in eating behavior and activity varied according to inter-generational relation
* Have a overview on the surgery as a turning point in the life of patients
* Estimate the relevant message of cares given to patients, in order to better adjust medical intervention, in conjunction with patients and their family members.

This is a prospective observational study. It will be performed in two university hospitals: CHU Ambroise Paré at Boulogne-Billancourt city and CHU Pitié Salpétrière at Paris, in nutrition department and metabolic surgery department. The study will involve collaboration of a team of social researchers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Eligible to undergo bariatric surgery
* Post bariatric surgery follow-up visits will take place in the nutrition department
* Living together with family member (children aged 11-17 years, parents, spouse, cohabitee or partner in civil union)
* Informed consent signed

Exclusion Criteria:

* Higher-order cognitive disorders
* Language difficulties in understanding
* Living alone or living without any family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo bariatric surgery (bypass or sleeve) and live together with their families.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in different eating habits and culinary items in responses to questionnaires | At 3 month, 6 month and 12 month
  Changes from baseline in different eating habits and culinary items in responses to questionnaires at 3 months, 6 months and 1 year after bariatric surgery. It is expected that patient's feeding practice should be in accordance with the postsurgical dietary guidelines.

SECONDARY OUTCOMES:
Changes from baseline in different items about physical activity in responses to questionnaires | At 3 month, 6 month and 12 month
  Changes from baseline in different items about physical activity in responses to questionnaires at 3 months, 6 months and 1 year after bariatric surgery. It is expected that patient's physical activity practice should be in accordance with the postsurgical guidelines.
Quality of life measured by scores | At baseline, 3 month, 6 month and 12 month
  Quality of life will be measured by scores at baseline, 3 month, 6 month and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Czernichow, MD, PhD, Principal Investigator — CHU Ambroise Paré; Kàtia Lurbe-Puerto, PhD, Study Director — CHU Ambroise Paré
Locations (1):
- Department of Nutrition, CHU Ambroise Paré, Boulogne-Billancourt, Hauts Des Seine, France